CLINICAL TRIAL: NCT00892749
Title: A Phase 3, Long-term Study in Patients With Chronic Kidney Disease (CKD) and Hyperphosphatemia on Hemodialysis
Brief Title: Long-term Study in Patients With Chronic Kidney Disease and Hyperphosphatemia on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1585-CL-0004
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease; Renal Dialysis; Renal Insufficiency; Hyperphosphatemia
Keywords: hyperphosphatemia; hemodialysis; CKD; ASP1585
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1. ASP1585 (Experimental)
  Interventions: Drug: ASP1585

INTERVENTIONS:
Drug: ASP1585 — oral
  Other Names: ILY101; AMG223

SUMMARY:
This is a multi-center, open-labeled, non-comparative study to examine the safety and efficacy of ASP1585 for long-term dosing in chronic kidney disease and hyperphosphatemia patients on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients on hemodialysis
* Hyperphosphatemia
* Written informed consent

Exclusion Criteria:

* Patients with gastrointestinal surgery or enterectomy
* Severe cardiac disease patients
* Patients with severe constipation or diarrhea
* Patients with a complication of malignant tumors
* Patients with uncontrolled hypertension
* Patients treated with parathyroid intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Changes in serum Phosphorus level | After 48 weeks

SECONDARY OUTCOMES:
Percent of the patients meeting the target range of serum Phosphorus levels | During the treatment
Changes in serum Calcium level | After 48 weeks
Changes in serum Ca x P | After 48 weeks
Changes in intact PTH level | After 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Chugoku
  - Chūbu
  - Kansai
  - Kantou